CLINICAL TRIAL: NCT04804111
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Dose-finding Phase 2b Clinical Trial to Evaluate the Efficacy and Safety of URC102 in Patient With Gout
Brief Title: Study of of URC102 to Assess the Efficacy and Safety in Gout Patients
Acronym: URC102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JWP-URC-203
Record Dates: First submitted 2020-11-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-11

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): maintain the initial dose, without increasing the dose.
  Interventions: Drug: arm 0
- URC102 3mg (Active Comparator): Administer 3 mg of URC102 for 12 weeks
  Interventions: Drug: arm 1
- URC102 6mg (Active Comparator): Administer 3 mg of URC102 for 1 week and 6 mg of URC102 for 11 Weeks.
  Interventions: Drug: arm 2
- URC102 9mg (Active Comparator): Administer 3 mg of URC102 for 1 week and 6 mg of URC102 for 1 Weeks, maintain 9 mg of URC102 dose
  Interventions: Drug: arm 3
- Febuxostat 80 mg (Other): maintain the initial dose, without increasing the dose.
  Interventions: Drug: arm 4

INTERVENTIONS:
Drug: arm 0 — placebo group
  Arms: Placebo
Drug: arm 1 — 3 mg of the URC102 group
  Arms: URC102 3mg
Drug: arm 2 — 6 mg of the URC102 group
  Arms: URC102 6mg
Drug: arm 3 — 9 mg of the URC102 group
  Arms: URC102 9mg
Drug: arm 4 — Febuxostat 80 mg
  Arms: Febuxostat 80 mg

SUMMARY:
To confirm the safety and efficacy (dose response and optimal dose according to the serum uric acid response rate) of URC102 when orally-administered to patients with gout and gout-related hyperuricemia in comparison with placebo.

Therapeutic dose-finding study, Placebo-controlled, randomized, double-blind, multicenter, phase 2 clinical trial.

DETAILED DESCRIPTION:
Placebo-controlled, randomized, double-blind, multicenter, phase 2 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Screening Inclusion Criteria The subjects must meet all the following criteria to be eligible for articipation in this study.

  1. Subjects who are aged ≥19 and <70 years at the time of providing written informed consent
  2. Subjects who are diagnosed with gout according to American College of Rheumatology (1977) criteria for the classification of acute arthritis of primary gout.
  3. Subjects who have the ability and willingness to actively conduct TLC recommended in this study
  4. Subjects who provided written informed consent to voluntarily participate in the study
* Randomization Inclusion Criterion. Subjects who meet the screening inclusion criteria will be randomly assigned to the following criteria.

  1. sUA ≥ 7.0 mg/dL at Visit 2

     Exclusion Criteria:

  <!-- -->

  1. Subjects who have medical history or comorbidity as follow; (1) Active malignancy or history of malignancy within the past 5 years at the time of screening (2) Urolithiasis (3) Clinically important allergic disease (anaphylactic shock, etc.) (4) Lesch-Nyhan syndrome (5) Hereditary problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption (6) Ischemic heart diseases or congestive heart failure (7) Organ transplantation (recipient or scheduled to receipt)
  2. Subjects who have comorbidity or abnormality of lab results as follows; (1) Uncontrolled diabetes mellitus with drug therapy

     * HbA1c ≥ 9% or
     * Fasting plasma glucose (FPG) ≥160 mg/dL (2) Uncontrolled hypertension with treatment
     * Systolic blood pressure (SBP) ≥180 mmHg or
     * Diastolic blood pressure (DBP) ≥ 110 mmHg (3) Uncontrolled dyslipidemia with treatment
     * Total cholesterol ≥ 250 mg/dL (at least 8 hours of fasting) (4) Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 X upper limit of normal (ULN) or Total bilirubin ≥ 1.5 X ULN (5) eGFR* < 60 mL/min/1.73m2 * eGFR (MDRD equation) GFR(ml/min/1.73m2) = 186 × (SCr)-1.154 × (age)-0.203 × (0.742 if female) × (1.210 if African American) (6) Uncontrolled thyroid function with treatment (thyroid-stimulating hormone (TSH) ≥ 1.5 X UNL
  3. Subjects who are judged by the investigator to have a clinical cardiovascular disease that may affect the study based on the 12-lead ECG obtained at screening or those suspected to be at such risk
  4. Patients who have received or plan to receive any XOI or uricosuric agents within 3 weeks prior to study treatment
  5. Patients who have received or plan to receive diuretics or any medication action on human Uric Acid Transporter 1(hURAT1) such as indomethacin, pyrazinamide, fenofibrate, atorvastatin, amlodipine, losartan, captopril, enalapril, salicylates etc. within 2 weeks prior to study treatment However, those who have been on stable doses as below are allowed to participate in the study, if the administration method and dosage remain the same during the study period (1) Diuretics (thiazide only or thiazide-based combination, etc.) and antihypertensive agents (losartan etc.) used for the treatment of hypertension (2) Fenofibrate or lipid lowering drugs (atorvastatin) used for hyperlipidemia (3) Salicylates (aspirin)
  6. Patients who have been administered or plan to administer Mercaptopurine, Azathioprine, Theophyline within 1 week or within more than 5 times of its half-life prior to the Visit 1
  7. HIV Ag/Ab, HBs Ag or HCV Ab positive at screening
  8. Subjects who have known hypersensitivity or allergy to IPs (URC102 or febuxostat) or any components in their formulations
  9. Subjects who have childbearing or nursing
  10. Subjects who agree to use methods of birth control* during the study period and for up to 7 days after the final administration of the IP

      * Methods of birth control: ① intrauterine device or birth control implant, ② dual protection (condom with spermicide and contraceptive diaphragm or contraceptive sponge or cervical cap ③ surgical sterilization (vasectomy or tubal ligation or etc.)
  11. Subjects who have been administered any other IP or investigational device by participating in other studieswithin 4 weeks or within more than 5 times of its halflife prior to the Visit 1
  12. Subjects who have a history of drug or alcohol abuse within 5 years prior to the Visit 1
  13. Subjects who have any other reason that may affect the study or those who are judged by the investigator to be ineligible for participation in the study

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Serum uric acid response rate (< 6.0 mg/dL) at week 4 after the IP administration. | Week 4

SECONDARY OUTCOMES:
Serum uric acid response rate (< 5.0 mg/dL) at week 4 after the IP administration. | Week 4
Percent Change in Serum Uric Acid from Baseline to week 4 | Week 4
Change in Serum Uric Acid at week 4 from Baseline | Week 4
The Incidence rate of gout attack from baseline to week 4 | week 4
Serum uric acid response rate(< 6.0 mg/dL) at week 8 and week 12 after the IP administration | Week 8, Week 12
serum uric acid response rate(< 5.0 mg/dL) at week 8 and week 12 after the IP administration | Week 8, Week 12
Percent Change in Serum Uric Acid from Baseline to week 8 and week 12 | Week 8, Week 12
Change in Serum Uric Acid at week 8 and 12 from Baseline | Week 8, Week 12
The Incidence rate of gout attack from baseline to week 8 and 12 | Week 8, Week 12

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - JW Pharmaceutical, Seoul
  - Chung-Ang University Hospital, Seoul

REFERENCES:
- [Derived] Jun JB, Lee HS, Kim SH, Lee SG, Lim DH, Kim J, Park YB, Lim MJ, Hong SJ, Choi HJ, Lee SS, Kim HA, Hwang J, Suh CH, Han S, Choe JY, Yoo WH, Song JS. Efficacy and safety of epaminurad, a potent hURAT1 inhibitor, in patients with gout: a randomized, placebo-controlled, dose-finding study. Arthritis Res Ther. 2025 May 26;27(1):113. doi: 10.1186/s13075-025-03577-w. PMID 40420308